CLINICAL TRIAL: NCT06752174
Title: A Randomized, Blinded, Parallel Positive-controlled Clinical Trial of Sequential Vaccination of Sabin Inactivated Poliomyelitis Vaccine (Vero Cell) and Live Attenuated Poliomyelitis Vaccine in Healthy 2-month-old Infants
Brief Title: A Study to Evaluate Safety and Immunogenicity of Sequential Vaccination of Sabin Inactivated Poliomyelitis Vaccine (Vero Cell) and Live Attenuated Poliomyelitis Vaccine in Healthy 2-month-old Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017L00935-2
Record Dates: First submitted 2024-12-12; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Poliomyelitis
Keywords: sIPV; bOPV; sequential immune
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): study group: sIPV-sIPV-bOPV, a total of 3 doses, with 1 month between each vaccination; 150 participants
  Interventions: Biological: sIPV+bOPV
- control group (Active Comparator): control group: wIPV-wIPV-bOPV, a total of 3 doses, with 1 month between each vaccination; 150 participants
  Interventions: Biological: wIPV+bOPV

INTERVENTIONS:
Biological: sIPV+bOPV — 2+1 sequential" immunization program (sIPV-sIPV-bOPV)
  Arms: study group
Biological: wIPV+bOPV — 2+1 sequential" immunization program (wIPV-wIPV-bOPV)
  Arms: control group

SUMMARY:
The goal of this clinical trial is to evaluate the immunogenicity and safety of a Sabin Inactivated Poliomyelitis Vaccine (sIPV) and a commercially available Live Attenuated Poliomyelitis Vaccine (bOPV) according to the "2+1 sequential" immunization program (sIPV-sIPV-bOPV) in 2-month-old healthy infants.

DETAILED DESCRIPTION:
A total of approximately 300 infants 2 months of age (over 60 days old and less than 90 days old) will be enrolled and randomized in 1:1 ratio into the study group and control group, with 150 participants in each group.The study group will receive study sIPV developed by Biominhai and control group will receive wIPV developed by SANOFI PASTEUR S.A. The "2+1 sequential" procedure consists of 2 doses of inactivated vaccine (sIPV or wIPV) and 1 dose of bOPV, a total of 3 doses, with 1 month between each vaccination. This study has indicated that the sIPV is not inferior to the wIPV in terms of immunogenicity and safety according to the "2+1 sequential" immunization program in 2-month-old healthy infants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy permanent residents aged 2 months (over 60 days and less than 90 days);
2. Infant's legal guardians agree to sign the informed consent forms voluntarily;
3. Infant's legal guardians are able to comply with the requirements of the clinical trial protocol;
4. Armpit temperature ≤ 37.0 ℃

Exclusion Criteria:

1. Preterm birth (delivery before the 37th week of pregnancy).
2. Previous vaccination against polio.
3. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
4. History of polio.
5. History or family history of convulsions, seizures, encephalopathy, and neurological disorder.
6. History of a serious reaction to any prior vaccination or known hypersensitivity to any component of the investigational vaccine.
7. Individuals with immunodeficiency or receiving immunosuppression therapy.
8. Disturbance of coagulation diagnosed by doctor (e.g., coagulation factors deficiency, coagulation disease, platelet abnormality) or obvious bruising or coagulation disorder.
9. Known or suspected concomitant diseases include: respiratory disease, acute infection or active chronic disease, cardiovascular disease, liver and kidney disease, skin disease, mother with HIV infection.
10. Administration of blood or blood-related products or immunoglobulins (hepatitis B immunoglobulins is acceptable).
11. History of administration of live attenuated vaccines within 14 days.
12. History of administration of subunit or inactivated vaccines within 7 days.
13. Individuals with any acute diseases within 7 days, receiving antibiotics or antiviral therapy.
14. Fever within 3 days (Armpit temperature ≥38.0 ℃).
15. Use of any investigational product recently, or have any conditions that the investigator believes may affect the evaluation of the trial.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
The positive seroconversion rates of poliovirus type I, type II and type III neutralizing antibody | Day 30 post full vaccination

SECONDARY OUTCOMES:
GMT of poliovirus type I, type II and type III neutralizing antibody | Day 30 post full vaccination
GMI of poliovirus type I, type II and type III neutralizing antibody | Day 30 post full vaccination
The seropositive rates of poliovirus type I, type II and type III neutralizing antibody | Day 30 post full vaccination
The ratio of poliovirus type I, type II and type III neutralizing antibody titer ≥1:64 | Day 30 post full vaccination
Incidence of adverse reactions/events | 30 days after each dose of vaccination
Incidence of serious adverse events (SAE) | From the first immunization to 6 months after the last immunization

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Center for Diseases Control and Prevention, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No